CLINICAL TRIAL: NCT00097513
Title: National Cooperative Growth Study (NCGS) of Optimal Nutropin AQ and Nutropin Dosing in Pubertal Growth Hormone-Deficient (GHD) Subjects
Brief Title: National Cooperative Growth Study (NCGS) of Optimal Nutropin AQ and Nutropin Dosing in Pubertal Growth Hormone-Deficient (GHD) Patients
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Disclosures Group, Genentech, Inc.
Other Study IDs: 85-036, Substudy 12
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Dwarfism, Pituitary
Keywords: Pubertal Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is a multicenter, open-label, observational, postmarketing surveillance study that will collect information on the use of Genentech GH preparations to treat GH-deficient subjects with optimal GH dosing during puberty.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent boys who are GH deficient and Tanner Stage 2 or greater (testes 3 mL or greater)
* Adolescent girls who are GH deficient and breast Tanner Stage 2 or greater
* Current treatment with GH dose of 0.4 to 0.7 mg/kg/wk
* Ability to keep follow-up appointments throughout the study
* Willingness to remain on therapy until epiphyseal closure is achieved
* Prior enrollment in NCGS Core Study 85-036

Exclusion Criteria:

* Treatment with non-Genentech GH preparation
* Closed epiphyses
* Active neoplasia
* Treatment with insulin for diabetes

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pubertal Growth Hormone Deficiency
Sampling Method: Probability Sample
Dates: Start 2003-02; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lippe, M.D., Study Director — Genentech, Inc.
Locations (1):
- Genentech Central Contact, South San Francisco, California, United States